CLINICAL TRIAL: NCT00826566
Title: Pilot Study to Investigate the Anti-inflammatory Effects of Caffeine in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Anti-inflammatory Effects of Caffeine in Chronic Obstructive Pulmonary Disease (COPD) Subjects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Suitable subjects could not be recruited within the estimated time frame.
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Technologiestichting STW (NWO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STW6041
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; caffeine; chronic systemic inflammation; oxidative stress; supplementation; stable COPD GOLD stage II with CRP levels ≥ 3 mg/l
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 500 mg caffeine capsules per day
  Interventions: Dietary Supplement: Caffeine
- 2 (Placebo Comparator): 500 mg placebo capsules
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — 2 times 250 mg caffeine per day
  Arms: 1
Dietary Supplement: placebo — 2 times 250 mg per day
  Arms: 2

SUMMARY:
Nowadays it has become evident that a chronic systemic inflammation is present in patients suffering from chronic obstructive pulmonary disease (COPD).

The role of the nuclear enzyme poly(adenosine diphosphate-ribose)polymerase (PARP) as a key mediator within these systemic inflammatory processes as well as in COPD associated exercise intolerance and muscle weakness could recently been identified. The attenuating effect of dietary ingredients with PARP inhibiting activity on systemic inflammation was supported by data from in vitro and in vivo studies, from other groups as well as from our own lab. We identified several caffeine metabolites as potent inhibitors of the most abundant PARP-isoform PARP-1 in-vitro, in animal models as well as in ex-vivo experiments with whole blood from COPD patients.

However, clinical data with respect to their anti-inflammatory effects in COPD patients are currently not available for none of these substances. Therefore, the current clinical pilot study is intended to establish for the first time clinical data (proof of principle) on the anti-inflammatory potential of caffeine metabolites.

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD stage II (50% ≤ FEV1< 80%)
* CRP plasma levels ≥ 3 mg/l
* BMI > 20 kg/m2 and < 30 kg/m2
* Diastolic blood pressure (DBP)=60-90 mmHg, Systolic blood pressure (SBP)=100 150 mmHg

Exclusion Criteria:

* Physical and/or mental disease or major surgery in the present or the past that might limit participation in or completion of the study
* Reported current or previous metabolic (e.g. diabetes), cardiovascular and/or renal diseases
* Known presence of a carcinoma
* Acute and/or chronic inflammatory condition such as arthritis, arthrosis, chronic colitis, etc. during three months before entry of the study
* Respiratory tract infection or exacerbation of COPD for at least 8 weeks prior to the start of the study
* Change in treatment regime of the COPD subjects for at least 8 weeks prior to the start of the study
* Use of laxatives, anti-diarrhoeal drugs and any other medication that can influence the uptake of the investigational products and/or influence their metabolism during the trial
* During the month prior to the start of the study and during the study the use of antibiotics and/or local and systemic steroidal (glucocorticoids) and non-steroidal anti-inflammatory drugs (NSAID)
* Abnormal constant dietary eating habits and a coffee consumption of less than 3 cups per day (i.e. a usual daily intake of <400 mg caffeine).

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of C-reactive protein (CRP) and the cytokines TNF-a, IL-6, IL-8 and IL-10. | at the start and at the end of the intervention periods

SECONDARY OUTCOMES:
Activation of poly-(ADP-ribose) polymerase (PARP)-1 activation and DNA repair in peripheral lymphocytes | at the start and the end of the intervention periods
Oxidative stress markers in plasma such as PGF2alpha | at the start and the end of the intervention periods
Plasma concentrations of caffeine and metabolites | at the start and the end of the interventions
Gene transcription levels of cytokines, redox enzymes and other proteins involved in inflammatory and oxidative stress response | at the start and the end of the interventions
Cytokine concentrations in whole blood after ex vivo stimulation with LPS | at the start and the end of the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Geja J Hageman, PhD, Principal Investigator — Dept. of Health Risk Analysis and Toxicology, UMC+, Maastricht, The Netherlands; Antje R Weseler, PhD, Principal Investigator — Dept. of Pharmacology & Toxicology, UMC+, Maastricht, The Netherlands; Aalt Bast, PhD, Prof., Study Director — Dept. of Pharmacology & Toxicology, UMC+, Maastricht, The Netherlands
Locations (1):
- Maastricht University Medical Centre (UMC+), Maastricht, Netherlands